CLINICAL TRIAL: NCT03634839
Title: Effects of E-cigarette Flavors on Youth
Brief Title: Effects of E-cigarette Flavors on Youth TCORS 2.0
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2000023077-1; 2U54DA036151-06 (NIH)
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Nicotine Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Flavoring Agents; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Flavor and nicotine concentration is blinded to participant. Research staff and investigators are blinded to flavor order administer to participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sweet non-menthol, nicotine 36mg/ml (Experimental): Sweet flavor non-menthol (Watermelon) with 36mg/ml Nicotine
  Interventions: Drug: Flavoring Agents; Drug: Nicotine
- Sweet menthol, nicotine 36mg/ml (Experimental): Sweet flavor with menthol (Watermelon-menthol) with 36mg/ml Nicotine
  Interventions: Drug: Flavoring Agents; Drug: Nicotine

INTERVENTIONS:
Drug: Flavoring Agents — Flavor of e-liquid - sweet or tobacco
  Other Names: Cooling flavor
Drug: Nicotine — Nicotine level (36 mg/ml)
  Other Names: Nicotine concentration

SUMMARY:
This study is an examination of the influence of sweet and cooling flavors on the appeal and abuse potential of nicotine-containing e-cigarettes among susceptible youth.

DETAILED DESCRIPTION:
Researchers will examine the influence of sweet and cooling flavors on the appeal and abuse potential of nicotine-containing e-cigarettes among susceptible youth. Participants will rate the flavor intensity, coolness, sweetness, and irritation experienced using validated rating scales. Forty youth (18-20 years of age) who have experience with e-cigarettes and will participate in 1 laboratory session. They will receive 1 nicotine concentrations (36mg/ml nicotine salt) during the session; during the session they will be exposed, in random order, to sweet (watermelon) and sweet-cooling (watermelon-menthol) flavors combined with the assigned session nicotine concentration.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-20 years
* Able to read and write
* Used e-cigs at least 10 times in lifetime
* Used e-cigs in past 30 days

Exclusion Criteria:

* Current use of non-prescription substances besides nicotine, marijuana, alcohol
* Any significant current medical or psychiatric condition
* Known hypersensitivity to propylene glycol
* Pregnant or lactating females
* Uncontrolled asthma
* Nut/e-liquid flavorant allergy
* current marijuana (tetrahydrocannabinol) vaping + E-cigarette or vaping use Associated Lung Injury (EVALI) symptoms

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra Krishnan-Sarin, PhD, Principal Investigator — Yale University
Locations (1):
- CMHC, Substance Abuse Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Lim J, Wood A, Green BG. Derivation and evaluation of a labeled hedonic scale. Chem Senses. 2009 Nov;34(9):739-51. doi: 10.1093/chemse/bjp054. PMID 19833660
- [Derived] Li W, Davis DR, Wu R, Gueorguieva R, Green BG, Krishnan-Sarin S. The effect of "ice" components in sweet-flavored nicotine-containing e-liquids among young adult e-cigarette users. Exp Clin Psychopharmacol. 2025 Oct;33(5):477-482. doi: 10.1037/pha0000786. Epub 2025 Jun 9. PMID 40489161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 young adults (18-20 years) were screened for eligibility between November 7, 2022 and June 12, 2023 through Snapchat and referrals from previous participants.
Pre-assignment Details: A total of 40 participants completed the study. Specifically, 49 out of 84 participants were randomized, but 7 did not show up and 2 withdrew. Of the 35 who were not randomized, 18 did not meet inclusion criteria and 17 did not show up.
Groups:
- Sweet Non-menthol Then Sweet Menthol, Each With Nicotine 36mg/ml: Participants attended a one-time, two-hour laboratory session with two exposures to flavored nicotine-containing e-liquids in a randomized order. They first received Durasmoke watermelon (50:50 PG/VG base) e-liquid. After a 30-minute break, they then received Durasmoke watermelon-menthol (50:50 PG/VG base) e-liquid, each with a nicotine salt concentration of 36 mg/mL.
  Flavoring Agents: Flavor of e-liquid - sweet or tobacco
  Nicotine: Nicotine level (36 mg/ml)
- Sweet Menthol Then Sweet Non-menthol, Each With Nicotine 36mg/ml: Participants attended a one-time, two-hour laboratory session with two exposures to flavored nicotine-containing e-liquids in a randomized order. They first received Durasmoke watermelon-menthol (50:50 PG/VG base) e-liquid. After a 30-minute break, they then received Durasmoke watermelon (50:50 PG/VG base) e-liquid, each with a nicotine salt concentration of 36 mg/mL.
  Flavoring Agents: Flavor of e-liquid - sweet or tobacco
  Nicotine: Nicotine level (36 mg/ml)
Period: First Intervention (2 Hours)
Arm/Group | Sweet Non-menthol Then Sweet Menthol, Each With Nicotine 36mg/ml | Sweet Menthol Then Sweet Non-menthol, Each With Nicotine 36mg/ml
Started | 20 | 22
Completed | 20 | 20
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: 30 Minutes Break
Arm/Group | Sweet Non-menthol Then Sweet Menthol, Each With Nicotine 36mg/ml | Sweet Menthol Then Sweet Non-menthol, Each With Nicotine 36mg/ml
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Intervention (2 Hours)
Arm/Group | Sweet Non-menthol Then Sweet Menthol, Each With Nicotine 36mg/ml | Sweet Menthol Then Sweet Non-menthol, Each With Nicotine 36mg/ml
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sweet Non-menthol Then Sweet Menthol, Each With Nicotine 36mg/ml | Sweet Menthol Then Sweet Non-menthol, Each With Nicotine 36mg/ml | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.0 (0.7) | 19.2 (0.8) | 19.1 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 9 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 11 | 18 | 29
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
Currently enrolled in a degree program [Count of Participants; unit: Participants] | 17 | 15 | 32
Grade [Count of Participants; unit: Participants]
  Excellent (A's) | 14 | 13 | 27
  Good (B's) | 5 | 6 | 11
  Fair (C's) | 1 | 2 | 3
  Barely passing (D's) | 0 | 1 | 1
Preferred e-cigarette device [Count of Participants; unit: Participants]
  Disposable pod device | 16 | 20 | 36
  JUUL | 1 | 1 | 2
  Vape pen | 1 | 0 | 1
  Any pod device other than a JUUL | 2 | 1 | 3
Preferred e-cigarette nicotine level [Count of Participants; unit: Participants]
  50-59mg/mL or 5.0-5.9% | 14 | 16 | 30
  Other concentrations | 4 | 1 | 5
  I don't know the concentration | 2 | 5 | 7
Ever vaped cooling flavor [Count of Participants; unit: Participants] | 20 | 22 | 42
Past-month other tobacco use [Count of Participants; unit: Participants] | 12 | 12 | 24
Past-month vaped THC [Count of Participants; unit: Participants] | 18 | 7 | 25
Vaping age of onset [Mean (Standard Deviation); unit: years] | 14.8 (1.9) | 15.6 (1.7) | 15.2 (1.8)
Vaping frequency [Mean (Standard Deviation); unit: days per week] | 6.0 (1.8) | 6.1 (1.4) | 6.1 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Liking: Difference Score in Liking/Wanting of Each E-cigarette Condition
Description: The Labeled Hedonic Scale will be used to ask about liking and wanting of the e-cigarette (one item Visual Analog Scale with ratings ranging from "most disliked sensation imaginable" to "most liked sensation imaginable" with higher values indicating greater liking). Specific scale semantic structure and corresponding values: most disliked imaginable=-100, dislike extremely=-62.9, dislike very much=-41.6, dislike moderately=-17.6, dislike slightly=-5.9, neutral=0, like slightly=6.3, like moderately=17.8, like very much=44.4, like extremely=65.7, most liked imaginable=100.
Time Frame: Following administration of e-cigarette condition 1 (+10 minutes), following administration of e-cigarette condition 2 (+40)
Population: After each of the two puff bouts, we evaluated participants' reference for the overall experience of the e-cigarette using the LHS, which is a bipolar category ratio scale that spans from -100 (most disliked) to 100 (most liked), with 'neither liked nor disliked' positioned as the midpoint. The scale labels were places along the scale based on their semantic magnitude.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sweet Non-menthol, Nicotine 36mg/ml | Sweet Menthol, Nicotine 36mg/ml
Number analyzed (Participants) | 40 | 40
score on a scale | 1.268 (3.158) | -3.916 (3.158)
Statistical Analysis 1: Comparison: Sweet Non-menthol, Nicotine 36mg/ml vs Sweet Menthol, Nicotine 36mg/ml; Test type: Superiority; p = 0.053, t-test, 2 sided; Mean Difference (Final Values) = -5.184

2. Primary Outcome: Reinforcing Efficacy: Difference Score in Drug Effects of Each E-cigarette Condition
Description: Difference between e-cigarette effects for each e-cigarette condition as measured by the computerized version of the Drug Effects Questionnaire (DEQ). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. A modified version of the Drug Effects Questionnaire (DEQ) will be used in which participants rate acute responses to the e-cigarette on a 0-100mm scale from "not at all" (0mm) to "extremely" (100mm). Higher values indicate stronger reinforcing efficacy (i.e., wanting/liking effects).
Time Frame: as for outcome 1
Population: To examine wanting/liking, we used subscales from the Drug Effects Questionnaire (DEQ), following the approach established in previous literature. Four items were used to measure wanting/liking effects (the average of 'I feel good e-cigarette effects', 'I want more of that e-cigarette I received', 'I feel the e-cigarette strength', and 'I like the e-cigarette effect').
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sweet Non-menthol, Nicotine 36mg/ml | Sweet Menthol, Nicotine 36mg/ml
Number analyzed (Participants) | 40 | 40
score on a scale | 37.06 (3.01) | 35.18 (3.01)
Statistical Analysis 1: Comparison: Sweet Non-menthol, Nicotine 36mg/ml vs Sweet Menthol, Nicotine 36mg/ml; Outcome analyses will be intent-to-treat and using mixed-effects models with flavor as a within-subject factor. A significant main effect of flavor with greater liking of sweet plus cooling flavor than sweet minus cooling flavor will be considered supportive of our hypotheses; Test type: Superiority; p = 0.187, t-test, 2 sided; Mean Difference (Final Values) = -1.881

3. Primary Outcome: Craving: Change in Craving Score for E-cigarette
Description: Difference from baseline in craving for each e-cigarette condition will be measured by the Generalized Labeled Magnitude Scale (gLMS). Participants will self-report their craving for e-cigarettes using a computer mouse to indicate where on the scale response falls. The Generalized Labeled Magnitude Scales (gLMS) are category ratio scales with seven semantic labels: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable", positioned quasi-logarithmically as per empirically determined semantic magnitudes on a 0-100 scale (strongest imaginable at the 100 end).
Time Frame: At baseline (+0 minutes), Following administration of e-cigarette condition 1 (+10 minutes), following administration of e-cigarette condition 2 (+40)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sweet Non-menthol, Nicotine 36mg/ml | Sweet Menthol, Nicotine 36mg/ml
Number analyzed (Participants) | 40 | 40
score on a scale | 2.72 (0.22) | 2.43 (0.22)
Statistical Analysis 1: Comparison: Sweet Non-menthol, Nicotine 36mg/ml vs Sweet Menthol, Nicotine 36mg/ml; Test type: Superiority; p = 0.135, t-test, 2 sided; Mean Difference (Final Values) = -0.286

4. Primary Outcome: Irritation/Harshness: Difference Score in Irritation of Harshness of Each E-cigarette Condition
Description: Difference in irritation at each e-cigarette condition as measured by the computerized Generalized Labeled Magnitude Scale (gLMS). Participants will self-report their responses using a computer mouse to indicate where on the scale response falls. The Generalized Labeled Magnitude Scales (gLMS) are category ratio scales with seven semantic labels: "no sensation", "barely detectable", "weak", "moderate", "strong", "very strong", and "strongest imaginable", positioned quasi-logarithmically as per empirically determined semantic magnitudes on a 0-100 scale (strongest imaginable at the 100 end).
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Sweet Non-menthol, Nicotine 36mg/ml | Sweet Menthol, Nicotine 36mg/ml
Number analyzed (Participants) | 40 | 40
score on a scale | 20.92 (1.68) | 22.86 (1.68)
Statistical Analysis 1: Comparison: Sweet Non-menthol, Nicotine 36mg/ml vs Sweet Menthol, Nicotine 36mg/ml; Test type: Superiority; p = 0.210, t-test, 2 sided; Mean Difference (Final Values) = 1.942

ADVERSE EVENTS:
Time Frame: Two hours during a single lab session
Description: Two mild levels of adverse events were observed. The adverse event definition aligns with the definitions on ClinicalTrials.gov.
Groups:
- Sweet Non-menthol With Nicotine 36mg/ml: Participants attended a one-time, two-hour laboratory session with two exposures to flavored nicotine-containing e-liquids in a randomized order. They received Durasmoke watermelon (50:50 PG/VG base) e-liquid.
  Flavoring Agents: Flavor of e-liquid - sweet or tobacco
  Nicotine: Nicotine level (36 mg/ml)
- Sweet Menthol With Nicotine 36mg/ml: Participants attended a one-time, two-hour laboratory session with two exposures to flavored nicotine-containing e-liquids in a randomized order. They received Durasmoke watermelon-menthol (50:50 PG/VG base) e-liquid.
  Flavoring Agents: Flavor of e-liquid - sweet or tobacco
  Nicotine: Nicotine level (36 mg/ml)
Arm/Group | Sweet Non-menthol With Nicotine 36mg/ml | Sweet Menthol With Nicotine 36mg/ml
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 0/40 | 2/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sweet Non-menthol With Nicotine 36mg/ml (N=40) | Sweet Menthol With Nicotine 36mg/ml (N=42)
Vomiting (Product Issues) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT03634839/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT03634839/ICF_002.pdf